CLINICAL TRIAL: NCT06649214
Title: A Randomized, Double-blind, Double-dummy, Positive Drug Parallel Controlled Phase III Clinical Study to Evaluate the Safety and Efficacy of Olanzapine-Samidorphan Tablets in Adults With Schizophrenia
Brief Title: A Study of Olanzapine-Samidorphan Tablets in Adults With Schizophrenia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLG1130-301
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olanzapine-samidorphan (Experimental)
  Interventions: Drug: Olanzapine-samidorphan；
- Olanzapine (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine-samidorphan； — orally once daily, tablet, 10mg/10mg、15mg/10mg or 20mg/10mg，duration of 24 weeks.
  Arms: Olanzapine-samidorphan
Drug: Olanzapine — orally once daily, tablet, 10mg、15mg or 20mg，duration of 24 weeks.
  Arms: Olanzapine

SUMMARY:
The goal of this [clinical trial] is to [evaluate the safety and efficacy of olanzapine-samidorphan tablets] in [adults with schizophrenia]. The main question[s] it aims to answer are:

* [question 1] Olanzapine-samidorphan significantly mitigate weight gain better than olanzapine.
* [question 2] Olanzapine- samidorphan and olanzapine have similar antipsychotic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is age 18 to 55 years, inclusive.
* Subject has a BMI of 18.0 to 30.0 kg/m2, inclusive.
* Subject meets the DSM-5 criteria for a primary diagnosis of schizophrenia.
* PANSS total score ≥ 70.

Exclusion Criteria:

* Diagnosis of schizoaffective disorder or bipolar I or II disorder, or current, untreated or unstable major depressive disorder, or any other psychiatric condition that could interfere with participation in the study.
* Subject poses a current suicide risk in the opinion of the investigator.
* Subject has inflammatory bowel disease or any other gastrointestinal disorder associated with weight loss, anorexia nervosa, or binge eating disorder.
* Subject has a history of diabetes.
* Subject has used olanzapine, clozapine, chlorpromazine, or thioridazine at any time during the 6 months prior to screening or long-acting injectable antipsychotic medication in the last 6 months.
* Subject has taken opioid agonists within the 14 days prior to screening and/or anticipates a need to take opioid medication during the study period, or has taken opioid antagonists within 60 days prior to screening.
* Subject is taking any weight loss agents or hypoglycemic agents at screening.
* Subject has had a surgical procedure for weight loss or is planning to have liposuction during the study.
* Subject has a clinically significant or unstable medical illness, condition, or disorder that would be anticipated to potentially compromise subject safety or adversely affect the evaluation of efficacy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 654 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in body weight at Week 24. | 24 weeks
Proportion of subjects with ≥10% weight gain at Week 24. | 24 weeks